CLINICAL TRIAL: NCT00910403
Title: A Prospective Multicenter, Study to Evaluate the Safety and Effectiveness of the Presbyopia Algorithm for Hyperopia and Hyperopic Astigmatism Using LASIK
Brief Title: Multicenter Evaluation of Safety and Effectiveness of Presbyopic LASIK for Hyperopes
Acronym: PresbyLASIK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Dr. Gerhard Youssefi / VP Research & Clinical Operations, Technolas PerfectVision
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Presbyopia; Hyperopia
Keywords: Presbyopia; LASIK; Hyperopes
MeSH Terms: conditions — Presbyopia; Hyperopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: LASIK — Excimer Laser Ablation using LASIK
  Other Names: PresbyLASIK

SUMMARY:
The Presbyopia Algorithm subject to this study has been specifically developed to prospectively generate a treatment file for the Technolas 217z100 laser that will provide Presbyopia correction among eyes with primary hyperopia or hyperopic astigmatism (distance correction). The treatment algorithm provides a bilateral, multifocal ablation with a center near addition, thereby allowing good focus over a range of object distances.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years old
* Subjects must read, understand, and sign an Informed Consent Form (ICF).
* Subjects must be willing and able to return for scheduled follow up visits.
* Subjects must be willing to have both eyes treated during the same visit.
* Subjects must have up to +4 diopters (D) of absolute spherical hyperopia (not spherical equivalent), with up to +2.5 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction in both eyes. The spherical equivalent must be no more than +5.25 D.
* Subjects must have presbyopia as determined by an age-related need for optical aid (> +1.50 D) for reading with their best distance correction.
* Subjects who are contact lens wearers must have gas permeable (GP) lenses discontinued for at least 3 weeks and soft lenses discontinued for at least 1 week prior to the preoperative evaluation in the eye to be treated. Contact lens wearers who wear their contact lenses for any amount of time between the preoperative baseline examination and the operative visit must not be treated.
* Corneal topography should be normal.
* Subjects who are contact lens wearers must have 2 central keratometry readings and 2 manifest subjective refractions taken preoperatively at least one week apart. The refraction values must not differ by more than 0.50D as defined by manifest refraction spherical equivalent (MRSE). The keratometry values must not differ from the previous values by more than 0.50D in either meridian.
* High contrast, manifest, best spectacle-corrected logMAR distance visual acuity (VA) must be correctable to at least 0.1 (20/25 or 6/7.5) in both eyes.

Exclusion Criteria:

* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively.
* Eyes for which the baseline manifest subjective refraction exhibits a difference of greater than 0.75D in sphere power, or a difference of greater than 0.50D in cylinder power, or a difference in cylinder axis of more than 15 degrees compared to the baseline cycloplegic subjective refraction. For manifest cylinder of less than 0.75D, the difference in cylinder axis will not be taken into consideration.
* Subjects for whom the preoperative assessment of the ocular topography indicates that one or both eyes are not suitable candidates for treatment based upon the suggested computer-simulated treatment plan.
* Any subject who is going to be co-managed by an ophthalmologist or optometrist who is not approved as a Technolas GmbH Excimer laser Investigator.
* Subjects with anterior segment pathology, including dry eye syndrome and cataracts which in the Investigator's opinion, would interfere with best spectacle-corrected VA (BSCVA) or a successful treatment.
* Subjects with evidence of retinal vascular disease.
* Subjects with any residual, recurrent, or active ocular disease, or corneal abnormality that in the Investigator's opinion would interfere with BSCVA or a successful treatment.
* Subjects with signs of keratoconus.
* Subjects with unstable central keratometry readings with irregular mires.
* Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of excimer laser surgery for either refractive or therapeutic purposes.
* Subjects who have a history of Herpes simplex or Herpes zoster keratitis.
* Subjects who have a history of glaucoma or glaucoma suspect.
* Subjects who are immunocompromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, diabetes, autoimmune diseases and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Subjects taking systemic medications likely to affect wound healing such as corticosteroids or antimetabolites.
* Subjects who are known to be pregnant, lactating, or who plan to become pregnant during the course of the study.
* Subjects with known sensitivity to medications used for standard LASIK.
* Subjects participating in any other ophthalmic clinical trials during this clinical trial.
* Subjects with an ocular muscle disorder including a strabismus or nystagmus, or other disorders affecting fixation.
* Subjects at risk for angle closure.

Exclusion Criteria-For Fellow (Second) Eyes in Simultaneous Bilateral Treatment

Procedures:

* Flap complications during the first eye's surgery such as a free cap, partial flap, thin flap, or irregular flap.
* Epithelial defect exceeding 2mm x 2mm in dimension, or clinically significant debris in the interface between the flap and underlying stroma for the first eye.
* Severe blepharospasm in the first eye that may have prevented or impeded the completion of the keratectomy and/or the laser ablation procedure.
* Poor subject cooperation with instructions for the first eye's surgery and/or poor subject fixation on the laser fixation target.
* Aborted LASIK procedure in the first eye or PRK or Epi-LASIK was performed in the first eye because LASIK was not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected VA better than 20/40 | 6 M

SECONDARY OUTCOMES:
Percentage of eyes within +/- 1D from target refraction | 6M

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Chaubard, Dr., Principal Investigator — VisionFuture / Nice
Locations (4):
- France (3):
  - Dr. Roure, Nice
  - Vision Future Nice, Nice
  - Clinique de la Vision Paris, Paris
- Instituo Oftalmologico Casteanera, Barcelona, Spain